



#### **Statistical Analysis Plan Checklist**

Double-Blind Randomized Phase II Trial of Carboplatin and Pemetrexed with or without OGX-427 in Patients with Previously Untreated Stage IV Non-Squamous-Non-Small-Cell Lung Cancer

(The Spruce Clinical Trial)

Sponsor: Sarah Cannon Research Institute (SCRI)

**Development Innovations** 

Study Drug: OGX-427

SCRI Protocol Number: LUN 229

Prepared By: SCRI Development Innovations (Innovations)

Final version 1.0, 21MAY2015 

Confidential



# Statistical Analysis Plan Checklist for Investigator Initiated Trials History of Changes

This document has undergone the following changes:

| Version | | |
|---|---|---|
| Number | Version Date | Description of Changes |
| Draft 1.0 | 15JUL2014 | Original document [Prepared by Bryan Lange] |
| Draft 2.0 | 14AUG2014 | Updated based on Dr. Kajdasz's comments [Prepared by Bryan Lange] |
| Draft 2.1 | 06FEB2015 | Edited and updated by Shuangli Guo |
| Draft 3.0 | 21MAY2015 | Added clinical benefit rate (CBR) Stratified PFS, OS, ORR and CBR with baseline ECOG performance Added an exploratory objective |
| Final 1.0 | 21MAY2015 | |

Final version 1.0, 21MAY2015 





| 1 Introduction | |
|---|---|
| 1.1 Objectives | |
| Primary Objective: | To compare the progression-free survival (PFS) of OGX-427 plus carboplatin/pemetrexed therapy versus placebo plus carboplatin/pemetrexed in previously untreated patients with advanced non-squamous NSCLC. |
| Secondary<br>Objectives: | <ul> <li>To compare the objective response rate (ORR) in each treatment arm.</li> <li>Objective response rate in a poor performance subgroup (prospectively defined in patients with a baseline ECOG 0 vs.1)</li> <li>To compare overall survival (OS) in each treatment arm.</li> <li>Overall survival in a poor performance subgroup (prospectively defined in patients with a baseline ECOG 0 vs.1)</li> <li>Progression-free survival in a poor performance subgroup (prospectively defined in patients with a baseline ECOG 0 vs.1)</li> <li>To evaluate safety.</li> <li>Correlative analyses of serum levels of Hsp27.</li> </ul> |
| Objectives: | <ul> <li>Correlative analysis of treatment outcomes with specific biomarkers.</li> <li>Based on the observations from primary analysis, post <i>ad hoc</i> prognostic statistical modeling will be performed, with survival as a function of multiple baseline covariates using proportional hazards regression. Selection of prognostic terms will be based on hierarchical step-down. Note: Interactions were appropriate may be used for inclusion in the model and models with continuous variables dichotomized at median will also be evaluated. Coefficients of the Control Arm model will be used (or carried forward) to compute a "statistical model" score for all patients in the study (both arms). Primary evaluation of the statistical model score will be based on dichotomization at overall median score for all study patients resulting in classifying patients as "poor" versus "good" prognosis.</li> </ul> |
| 1.2 Study Design | |
| Study Type | □ Non-Randomized □ Randomized (Allocation Ratio: 1:1) |
| Details | This is a randomized, double-blind, placebo-controlled, Phase II trial comparing pemetrexed and carboplatin plus OGX-427 followed by maintenance pemetrexed and OGX-427 versus pemetrexed and carboplatin plus placebo followed by maintenance pemetrexed and placebo in patients with previously untreated advanced non-squamous NSCLC. The patients, investigator, study team members, (except for the mixing pharmacist/nurse), and anyone involved with the conduct of the trial from the time of randomization until database lock for the primary endpoint analysis will be blinded to the identity of the treatment assignment (OGX-427 or placebo). The primary endpoint of the trial is PFS. A total of 155 patients will be randomized in a 1:1 ratio. Randomization will be stratified by histology (adenocarcinoma vs. large cell carcinoma) and smoking status (smoker vs. non- |
| | smoker) for the purpose of balance of enrollment and exploratory analysis. Progression-Free Survival Follow-Up |
| | Patients who discontinue trial treatment prior to the occurrence of disease progression will be followed every 6 weeks from the date of last dose of study drug until disease progression or |

Final version 1.0, 21MAY2015 

REFERENCE SOP: CDS-0102 Template ID: ASSOC-DOC-116-SOP [A] Confidential





Final version 1.0, 21MAY2015 





| | ☐ Independent DSM |
|---|---|
| | ☐ Annual Report |
| | Abstract / Scientific Presentation (Oral/Poster) |
| Final Analysis | The final analysis will be conducted when 117 progression-free survival events are observed out of approximately 155 randomized patients. |
| 1.5<br>Responsibilities | |
| Trial Statistician: | Prepare SAP (or SAP check list) and TFL shells |
| Shuangli Guo | Review deliverables produced by Statistical Programmer or other Biostatistician |
| | Prepare TFLs for abstract submission and meeting presentation |
| | Clinical review |
| | The final statistical analysis |
| PK Statistician: | Not applicable |
| Independent | Prepare randomization scheme |
| Statistician: | Un-blinded safety delivery review and interim un-blinded analysis |
| David Bass | Validate statistical analysis methods and TFLs output |
| 1.6 Analysis<br>Software | |
| Main statistical analysis: | SAS Version 9.3 or above |
| Other analysis software: | None |
| 1.7 Coding | |
| | ☑ MedDRA: ☐ Version 17.0 |
| ☐ Medical History | |
| | ⊠ NCI-CTCAE Version 4.03 |
| □ Concomitant | ⊠ WHO-Drug: ☐ Version September 2014 |
| Medication | ☐ |
| ☐ Prior Therapy | |
| Subsequent/Further Therapy | |
| 3 Analysis<br>Population | |
| Intent-To-Treat | ☐ All patients who have started treatment in the study |
| (ITT) Population definition: Full | ☑ All patients who have been randomized in the study, regardless of whether they have |

Final version 1.0, 21MAY2015 



REFERENCE SOP: CDS-0102

LUN 229 Statistical Analysis Plan Checklist

| Analysis set | received any treatment or not All patients who have been randomized and have started treatment in the study Other definition, specify: |
|---|---|
| Per Protocol (PP)<br>Population to be<br>used in analysis: | ☐ Yes ☐ No If yes, please specify the criteria for exclusion from the PP population: |
| Safety (SAF)<br>Population<br>definition | <ul> <li>✓ All patients who have started treatment in the study. Patients will be analysed according to the actual treatment they have received.</li> <li>☐ Other definition, specify:</li> </ul> |
| Other Analysis Population definition: ECOG Performance Analysis set | A subset of the Full Analysis Set including only patients with a baseline ECOG ≤1 |
| 4 Baseline Value Definitions | |
| | The study-wise baseline value is defined as the most recent value prior to first study drug administration, and the cycle-wise baseline value is the most recent value prior to a given cycle's initial study drug administration. The clinical database has been designed such that both study-wise and cycle-wise baseline values are clearly identifiable and do not require derivation. |
| 5 Efficacy | |
| Response Criteria<br>Used: | □ RECIST 1.0 □ RECIST 1.1 □ Cheson 2007 □ Modified RECIST – specify: □ Other criteria, Specify: |
| Efficacy<br>Assessment<br>Timepoints: | Progression-free survival (PFS) and Objective response rate (ORR): Response to treatment will be evaluated every 6 weeks. Overall survival (OS): Survival will be followed from date of randomization to the date of death due to any cause, or the date the patient was known to be alive at the date of cutoff for the analysis. Schedule of assessments are tabulated in protocol Appendix D and descripted in section 7. |

Final version 1.0, 21MAY2015 





| Efficacy Endpoints: | | | |
|---|---|---|---|
| | | Endpoint | Primary Analysis Population |
| | Primary | Progression-free survival (PFS): death or disease progression via RECIST v1.1 | Full analysis set |
| | Secondary | Overall Survival (OS): death | Full analysis set |
| | | Objective Response Rate (ORR), Clinical Benefit Rate (CBR) | Full analysis set |
| | | Poor performance with OS, ORR, CBR, and PFS: The proportion of patients with a baseline ECOG 0 vs. 1 | ECOG Analysis Set<br>(a subset of FAS) |
| Definition of Terms: | | | |
| ⊠ Response | | | onse<br>weeks apart. |
| | □ Complete | Response + Partial Response + Stable Disease ≥ 6 m | nonths |
| | ☐ Complete<br>Disease (a | | weeks apart) + Stable |
| | Other crite | ria, specify: | |
| ⊠ Progression | Target Lesio | n Progressive Disease | |
| | smallest (nad study), or the | 6 increase in the sum of the diameters of target lesion:<br>ir) sum while on study (this includes the baseline sum<br>appearance of one or more new lesions. Requires no<br>ease of a minimum of 5 mm over sum. | if that is the smallest on |
| | Non-Target L | esion Progressive Disease | |
| | target lesions<br>progression" of<br>substantial wo | of one or more new lesions and/or unequivocal progres. When the patient also has measurable disease, to a on the basis of the non-target disease, there must be a presenting in non-target disease such that, even in present, the overall tumour burden has increased sufficiently | chieve "unequivocal<br>an overall level of<br>ence of SD or PR in the |
| | Clinical Prog | ression | |
| | health status | symptomatic deterioration that is defined as global or such that it requires discontinuation of trial treatment vase progression at that time. | |
| ⊠ Subsequent<br>Therapy | | nerapy (subsequent treatment) is defined as therapy the OGX-427/Placebo. This will be collected during follow | |
| ☐ Treatment | Not applicable | <del></del> | |

Final version 1.0, 21MAY2015 

REFERENCE SOP: CDS-0102 Template ID: ASSOC-DOC-116-SOP [A] Confidential



Confidential



| Failure | | | |
|---|---|---|---|
| Definition of<br>Endpoints: | Start Date: Date of Randomization Date of First Treatment End Date (specify for all pertinent endpoints): Progression-Free Survival: Event = Progression or Death | | |
| | Situation | Date of Event or<br>Censoring | Outcome |
| | No baseline assessment | Date of randomization | Censored |
| | Progression documented between scheduled visits | First date of evaluated overall response = PD | Event |
| | No progression | Date of last evaluable tumor assessment | Censored |
| | Treatment discontinuation for adverse event or other reason | Date of last evaluable tumor assessment | Censored |
| | Further anti-cancer therapy started | Start date of latest anti-<br>cancer therapy | Censored |
| | Death before first PD assessment | Date of death | Event |
| | Death before the next scheduled tumour assessment | Date of death | Event |
| | Death after one missed tumour assessment but before second missed tumour assessment | Date of death | Event |
| | Death after two or more missed tumour assessment | Date of last evaluable tumour assessment | Censored |
| | Patient experiencing symptomatic deterioration before RECIST PD | Date of clinical disease progression | Event |
| | Overall Survival: Event = Death | | |
| | Situation | Date of Event or<br>Censoring | Outcome |
| | Death | Date of death | Event |
| | Alive on date of data cut-off | Date of data cut-off | Censored |
| | Alive before date of data cut-off, but status unknown on date of data cut-off (e.g. lost to follow-up) | Date of last contact | Censored |
| | Withdrawal Informed Consent | Date of informed consent withdrawn | Censored |
| ○ Objective Response Rate ○ CRP ○ CRP | Default: Estimates of rates in each treatment arm confidence intervals using the method of Cloppe | | xact 95% |
| (ORR) | □ Difference in ORR & 95% confidence interval | between treatment arms | |
| ☐ Disease Control Rate (DCR) | ☑ Proportions of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) and not evaluable (NE) will be calculated. | | |
| | ☑ p-value, specify statistical test: Fisher's exact | test | |
| ☐ Clinical Benefit<br>Rate (CBR) | | | |

Final version 1.0, 21MAY2015 

REFERENCE SOP: CDS-0102 Template ID: ASSOC-DOC-116-SOP [A]





REFERENCE SOP: CDS-0102

| ☐ Time To<br>Progression (TTP) | |
|---|---|
| □ Progression-<br>Free Survival (PFS) | Other quartiles or percentages of survival required, specify: |
| ☑ Overall Survival | ☐ Hazard ratio and two-sided 95% confidence interval between treatment arms, un-stratified (PFS and OS) |
| (OS) | □ p-value, specify statistical test: the un-stratified log-rank test |
| ☐ Duration of Response | ☐ Hazard ratio & 95% confidence interval between treatment arms, stratified (specify stratification factor(s)): |
| ☐ Duration of<br>Stable Disease | p-value, specify statistical test: |
| ☐ Time To<br>Treatment Failure<br>(TTF) | |
| Other, Specify: | |
| 6 Safety | |
| Adverse Events | Definition of Adverse Event: any adverse event (AE) that starts or worsens after the start of the first dose of study treatment up to 30 days post last dose. |
| Laboratory Data | Data will be summarized by: |
| | ☐ H/L for all lab parameters |

Final version 1.0, 21MAY2015 



#### Tier 1 Study - Tables, Figures & Listings

| Standard TFLs | Standard TFLs | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| Table 1 | Patient disposition | □ Number of patients consented □ Number of patients randomized □ Number of patients treated □ Reason for treatment discontinuation □ Reason for end of study | All randomized patients |
| Table 2 | Demographic characteristics | □ Age: Mean, SD, Median, Min, Max □ Age group: Senior (>=65) Adult (<65) □ Sex □ Race □ Ethnicity □ ECOG □ Tobacco use | Full analysis set |
| Table 3 | Disease history | <ul> <li>☐ Histology</li> <li>☐ Disease staging at study entry</li> <li>☐ Time from initial pathological diagnosis to randomization</li> <li>☐ Time from most recent recurrence or progression to randomization</li> <li>☐ EGFR Mutation Status</li> <li>☐ ALK Translocation</li> <li>☐ Sites of Metastatic Disease</li> </ul> | Full analysis set |
| Table 4 | Prior therapies – Systemic,<br>Radiation, and Surgery | Specify prior therapies groups to be summarized: prior systemic therapy, prior radiation therapy, and prior surgery | Full analysis set |
| Table 5 | Lab parameters at baseline | Specify lab parameters: | Safety analysis set |
| | | Haematology: Haemoglobin, Haematocrit, Platelets, White Blood Cells, Neutrophils, Lymphocytes, and Monocytes | |
| | | <u>Chemistry</u> : Albumin, Calcium, Carbon<br>Dioxide, Chloride, Creatinine, Glucose,<br>Potassium, Sodium, Total Protein, and<br>Blood Urea Nitrogen | |
| | | Liver function tests: SGPT/ALT,<br>SGOT/AST, Alkaline Phosphatase, and<br>Total Bilirubin | |
| Table 6 | Time on treatment and exposure | Initial planned dose, Cumulative actual dose, Actual dose intensity, Planned dose intensity, Relative dose intensity (%), Duration, Number of cycles treatment and maintenance, Dose modifications | Safety analysis set |
| Table 7 | Progression-free survival | Number of events, Number of censor,<br>Kaplan-Meier estimates of Median PFS<br>[months (95% CI)] | Full analysis set [Safety analysis set will be used if >10% of |

Final version 1.0, 21MAY2015 





| andard TFL | S | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| | | Probability of events at: 6 months and 12 months Hazard ratio and 95% CI between treatment groups using Cox proportional hazards model P-value between arms using log-rank test | randomized patients d<br>not receive study<br>treatment)]<br>ECOG analysis set |
| Table 8 | Overall survival | Number of deaths, Number of censor, Kaplan-Meier curves with Median OS [months (95% CI)] Probability of events at: 6 months and 12 months Hazard ratio and 95% CI between treatment groups using Cox proportional hazards model P-value between arms using log-rank test | Full analysis set [Safety analysis set wibe used if >10% of randomized patients donot receive study treatment)] ECOG analysis set |
| Table 9 | Response rates | Best overall response: Complete response (CR), Partial response (PR), Stable disease (SD), RECIST progressive disease (rPD), Clinical progressive disease (cPD), Not evaluable (NE), Unknown Objective response rate (ORR) (CR + PR): ORR, 95% Confidence interval Clinical Benefit Rate (CBR) (CR + PR+SD≥6months): CBR, 95% Confidence interval | Full analysis set [Safety analysis set wi be used if >10% of randomized patients d not receive study treatment)] ECOG analysis set |
| Table 10 | AE overview | Number of patient with at least: adverse events, related adverse events, serious adverse events (SAEs), related SAEs, SAE leading to death, related SAE leading to death, AE leading to treatment discontinued, AE leading to treatment interrupted, AE leading to treatment held, AE leading to treatment held, AE leading to treatment reduced | Safety analysis set |
| Table 11 | Summary of adverse events | System organ class, Preferred term | Safety analysis set |
| Table 12 | Summary of adverse events by grade | System organ class, Preferred term, CTCAE grade | Safety analysis set |
| Table 13 | Summary of related adverse events | System organ class, Preferred term | Safety analysis set |

Final version 1.0, 21MAY2015 

REFERENCE SOP: CDS-0102 Template ID: ASSOC-DOC-116-SOP [A] Confidential





| Standard TFLs | Standard TFLs | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| Table 14 | Summary of related adverse events by grade | System organ class, Preferred term, CTCAE grade | Safety analysis set |
| Table 15 | Summary of adverse events leading to treatment discontinuation | Preferred term | Safety analysis set |
| Table 16 | Summary of adverse events leading to dose reduction | Preferred term | Safety analysis set |
| Table 17 | Summary of deaths | Reasons of deaths | Safety analysis set |
| Table 18 | Summary of lab<br>parameters (worst grade<br>post-baseline) | CTCAE grade at baseline and maximum shift post-baseline: Haematology: Haemoglobin, Haematocrit, Platelets, White blood cells, Neutrophils, Lymphocytes, and Monocytes Chemistry: Albumin, Calcium, Carbon dioxide, Chloride, Creatinine, Glucose, Potassium, Sodium, Total protein, and Blood urea nitrogen Liver function tests: SGPT/ALT, SGOT/AST, Alkaline phosphatase, and Total bilirubin | Safety analysis set |
| Table 19 | Summary of follow-up duration | Time (months) for randomization to death, lost to follow-up, or completion of 2 year survival follow-up, whichever comes first. | Full analysis set |
| Table 20 | Summary of serum Hsp27<br>change from baseline over<br>time | serum Hsp27 level at baseline and protocol timepoint, percentage change of serum Hsp27 level from baseline | FAS, with serum Hsp27 measurement |

| Figure No | Description | Variables/Analyses To Be Included | Population |
|---|---|---|---|
| Figure 1 | Progression-Free Survival | Timescale to be used on horizontal axis: | Full analysis set |
| | | ☐ Day ☐ Week ☐ Year | ECOG analysis set |
| Figure 2 | Overall Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Full analysis set ECOG analysis set |

Final version 1.0, 21MAY2015 

#### **LUN229 TOC of TFL shells**

| Fable 2 Demographic Characteristics Full analysis set Fable 3 Disease History Full analysis set Fable 4 Prior Therapy Full analysis set Fable 5.1 Laboratory Parameters at Baseline - Hematology Full analysis set Fable 5.2 Laboratory Parameters at Baseline - Blood Chemistry Full analysis set Fable 5.2 Laboratory Parameters at Baseline - Liver Function Test Full analysis set Fable 6.1 Dose Exposure - Carboplatin Full analysis set Fable 6.2 Dose Exposure - Pemetrexed Full analysis set Fable 6.3 Dose Exposure - Pemetrexed Full analysis set Fable 6.4 Treatment Modifications - Carboplatin Full analysis set Fable 6.5 Treatment Modifications - Pemetrexed Full analysis set Fable 6.6 Treatment Modifications - Pemetrexed Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival Full analysis set Fable 7.2 Progression-free Survival Full analysis set Fable 8.1 Overall Survival - Statified by Baseline ECOG Performance Full analysis set Fable 8.1 Overall Survival - Statified by Baseline ECOG Performance Full analysis set Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Full analysis set Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Full analysis set Fable 9.1 Adverse Events by System Organ Class and Preferred Term Safety analysis set Fable 11 Adverse Events by System Organ Class and Preferred Term Safety analysis set Fable 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Full analysis set Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set Treatment-related Adverse Events by System Organ Class, Preferred Term Safety analysis set Treatment-related Adverse Events by System Organ Class, Preferred Term Safety analysis set Treatment-related Adverse Events by | TFL No. | TLF Title | Analysis Set |
|---|---|---|---|
| Fable 3 Disease History Fable 4 Prior Therapy Fable 5.1 Laboratory Parameters at Baseline - Hematology Fable 5.2 Laboratory Parameters at Baseline - Blood Chemistry Fable 5.3 Laboratory Parameters at Baseline - Liver Function Test Fable 6.1 Dose Exposure - Carboplatin Fable 6.2 Dose Exposure - Carboplatin Fable 6.3 Dose Exposure - Pemetrexed Fable 6.3 Dose Exposure - Pemetrexed Fable 6.3 Dose Exposure - Pemetrexed Fable 6.4 Treatment Modifications - Carboplatin Fable 6.5 Treatment Modifications - Carboplatin Fable 6.6 Treatment Modifications - Pemetrexed Fable 6.6 Treatment Modifications - OGX-427 or Placebo Fable 6.6 Treatment Modifications - OGX-427 or Placebo Fable 7.1 Progression-free Survival Fable 7.2 Progression-free Survival - Statified by Baseline ECOG Performance Fable 8.1 Overall Survival - Stratified by Baseline ECOG Performance Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline Fable 10 Adverse Events by System Organ Class and Preferred Term Fable 11 Adverse Events by System Organ Class and Preferred Term Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported Fable 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Fable 15.1 Adverse Events Leading to | Table 1 | Patient Disposition | All enrolled patients |
| Fable 4 Prior Therapy Full analysis set Fable 5.1 Laboratory Parameters at Baseline - Hematology Full analysis set Fable 5.2 Laboratory Parameters at Baseline - Blood Chemistry Full analysis set Fable 5.3 Laboratory Parameters at Baseline - Liver Function Test Fable 6.1 Dose Exposure - Carboplatin Full analysis set Fable 6.2 Dose Exposure - Pemetrexed Full analysis set Fable 6.3 Dose Exposure - OGX-427 or Placebo Full analysis set Fable 6.4 Treatment Modifications - Carboplatin Full analysis set Fable 6.5 Treatment Modifications - Pemetrexed Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival Fable 7.2 Progression-free Survival Fable 8.1 Overall Survival Fable 8.2 Overall Survival - Statified by Baseline ECOG Performance Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Fable 11 Adverse Events Overview Safety analysis set Fable 12 Adverse Events by System Organ Class and Preferred Term Adverse Events Overview Safety analysis set Fable 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Fable 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Full analysis set Fable 15 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term and Maximum Reported Full Adverse Events Safety analysis set Fable 15 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Full Adverse Events Safety analysis set Fable 15 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Full Adverse Events Safety analysis set Full Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Full Adverse Events Safety analysis set Full Adve | Table 2 | Demographic Characteristics | Full analysis set |
| Fable 5.1 Laboratory Parameters at Baseline - Hematology Full analysis set Fable 5.2 Laboratory Parameters at Baseline - Blood Chemistry Full analysis set Fable 5.3 Laboratory Parameters at Baseline - Liver Function Test Full analysis set Fable 6.1 Dose Exposure - Carboplatin Full analysis set Fable 6.2 Dose Exposure - Pemetrexed Full analysis set Fable 6.3 Dose Exposure - Pemetrexed Full analysis set Fable 6.4 Treatment Modifications - Carboplatin Full analysis set Fable 6.5 Treatment Modifications - Carboplatin Full analysis set Fable 6.6 Treatment Modifications - Pemetrexed Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival Full analysis set Fable 7.2 Progression-free Survival - Statified by Baseline ECOG Performance ECOG analysis set Fable 8.1 Overall Survival - Stratified by Baseline ECOG Performance ECOG analysis set Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance ECOG analysis set Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Fable 10 Adverse Events Overview Safety analysis set ECOG Performance Fable 11 Adverse Events by System Organ Class and Preferred Term Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term and Maximum Reported Safety analysis set Safe | Table 3 | Disease History | Full analysis set |
| Table 5.2Laboratory Parameters at Baseline - Blood ChemistryFull analysis setTable 5.3Laboratory Parameters at Baseline - Liver Function TestFull analysis setTable 6.1Dose Exposure - CarboplatinFull analysis setTable 6.2Dose Exposure - PemetrexedFull analysis setTable 6.3Dose Exposure - OGX-427 or PlaceboFull analysis setTable 6.4Treatment Modifications - CarboplatinFull analysis setTable 6.5Treatment Modifications - PemetrexedFull analysis setTable 6.6Treatment Modifications - OGX-427 or PlaceboFull analysis setTable 7.1Progression-free SurvivalFull analysis setTable 7.2Progression-free Survival - Statified by Baseline ECOG PerformanceECOG analysis setTable 8.1Overall Survival - Stratified by Baseline ECOG PerformanceECOG analysis setTable 9.1Best Overall Response, Objective Response Rate, and Clinical Benefit RateFull analysis setTable 9.2Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by BaselineECOG analysis setTable 10Adverse Events OverviewSafety analysis setTable 11Adverse Events by System Organ Class and Preferred TermSafety analysis setTable 12Adverse Events by System Organ Class, Preferred Term and Maximum ReportedSafety analysis setTable 13Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum ReportedSafety analysis setTable 14Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum | Table 4 | Prior Therapy | Full analysis set |
| Table 5.3Laboratory Parameters at Baseline - Liver Function TestFull analysis setTable 6.1Dose Exposure - CarboplatinFull analysis setTable 6.2Dose Exposure - PemetrexedFull analysis setTable 6.3Dose Exposure - OGX-427 or PlaceboFull analysis setTable 6.4Treatment Modifications - CarboplatinFull analysis setTable 6.5Treatment Modifications - PemetrexedFull analysis setTable 6.6Treatment Modifications - OGX-427 or PlaceboFull analysis setTable 7.1Progression-free SurvivalFull analysis setTable 7.2Progression-free Survival - Statified by Baseline ECOG PerformanceECOG analysis setTable 8.1Overall Survival - Stratified by Baseline ECOG PerformanceECOG analysis setTable 9.2Best Overall Response, Objective Response Rate, and Clinical Benefit RateFull analysis setTable 9.2Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by BaselineECOG analysis setTable 10Adverse Events OverviewSafety analysis setTable 11Adverse Events by System Organ Class and Preferred TermSafety analysis setTable 12Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE GradeSafety analysis setTable 13Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum ReportedSafety analysis setTable 14Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum ReportedSafety analysis set | Table 5.1 | Laboratory Parameters at Baseline - Hematology | Full analysis set |
| Table 6.1 Dose Exposure - Carboplatin Full analysis set Table 6.2 Dose Exposure - Pemetrexed Full analysis set Table 6.3 Dose Exposure - OGX-427 or Placebo Full analysis set Table 6.4 Treatment Modifications - Carboplatin Full analysis set Table 6.5 Treatment Modifications - Pemetrexed Full analysis set Table 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Table 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Table 7.1 Progression-free Survival Table 7.2 Progression-free Survival - Statified by Baseline ECOG Performance ECOG analysis set Table 8.1 Overall Survival - Stratified by Baseline ECOG Performance ECOG analysis set Table 8.2 Overall Survival - Stratified by Baseline ECOG Performance Table 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Table 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Table 10 Adverse Events Overview Table 11 Adverse Events Dy System Organ Class and Preferred Term Table 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Table 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term | Table 5.2 | Laboratory Parameters at Baseline - Blood Chemistry | Full analysis set |
| Full analysis set Full analysi | Table 5.3 | Laboratory Parameters at Baseline - Liver Function Test | Full analysis set |
| Fable 6.3 Dose Exposure- OGX-427 or Placebo Full analysis set Fable 6.4 Treatment Modifications - Carboplatin Full analysis set Fable 6.5 Treatment Modifications - Pemetrexed Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival Full analysis set Fable 7.2 Progression-free Survival - Statified by Baseline ECOG Performance Fable 8.1 Overall Survival - Stratified by Baseline ECOG Performance Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 10 Adverse Events Overview Fable 11 Adverse Events by System Organ Class and Preferred Term Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set Fable 15.1 Safety analysis set | Table 6.1 | Dose Exposure - Carboplatin | Full analysis set |
| Treatment Modifications - Carboplatin Full analysis set Treatment Modifications - Pemetrexed Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival Full analysis set Fable 7.2 Progression-free Survival - Statified by Baseline ECOG Performance Full analysis set Fable 8.1 Overall Survival - Stratified by Baseline ECOG Performance Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Full a | Table 6.2 | Dose Exposure - Pemetrexed | Full analysis set |
| Treatment Modifications - Pemetrexed Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Treatment Modifications - OGX-427 or Placebo Full analysis set Fu | Table 6.3 | Dose Exposure- OGX-427 or Placebo | Full analysis set |
| Table 6.6 Treatment Modifications - OGX-427 or Placebo Full analysis set Fable 7.1 Progression-free Survival - Statified by Baseline ECOG Performance Full analysis set Full a | Table 6.4 | Treatment Modifications - Carboplatin | Full analysis set |
| Fable 7.1 Progression-free Survival Full analysis set Fable 7.2 Progression-free Survival - Statified by Baseline ECOG Performance Fable 8.1 Overall Survival Full analysis set Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Fable 10 Adverse Events Overview Fable 11 Adverse Events by System Organ Class and Preferred Term Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 13 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Fable 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Fable 15.1 Safety analysis set Fable 15.1 Safety analysis set Fable 15.1 Safety analysis set Fable 15.1 Safety analysis set | Table 6.5 | Treatment Modifications - Pemetrexed | Full analysis set |
| Progression-free Survival - Statified by Baseline ECOG Performance Fable 8.1 Overall Survival Full analysis set Full analysi | Table 6.6 | Treatment Modifications - OGX-427 or Placebo | Full analysis set |
| Fable 8.1 Overall Survival Overall Survival - Stratified by Baseline ECOG Performance Fable 8.2 Overall Survival - Stratified by Baseline ECOG Performance Fable 9.1 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Fable 9.2 Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Fable 10 Adverse Events Overview Fable 11 Adverse Events by System Organ Class and Preferred Term Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Fable 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Fable 15.1 Safety analysis set | Table 7.1 | Progression-free Survival | Full analysis set |
| Overall Survival - Stratified by Baseline ECOG Performance Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Full analysis set Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Fable 10 Adverse Events Overview Fable 11 Adverse Events by System Organ Class and Preferred Term Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Fable 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set CTCAE Grade Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 7.2 | Progression-free Survival - Statified by Baseline ECOG Performance | ECOG analysis set |
| Best Overall Response, Objective Response Rate, and Clinical Benefit Rate Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG Performance Adverse Events Overview Adverse Events by System Organ Class and Preferred Term Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Adverse Events by System Organ Class, Preferred Term Table 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 8.1 | Overall Survival | Full analysis set |
| Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG analysis set ECOG Performance Adverse Events Overview Adverse Events by System Organ Class and Preferred Term Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Table 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set Safety analysis set | Table 8.2 | Overall Survival - Stratified by Baseline ECOG Performance | ECOG analysis set |
| ECOG Performance Fable 10 Adverse Events Overview Safety analysis set Fable 11 Adverse Events by System Organ Class and Preferred Term Safety analysis set Fable 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Safety analysis set Fable 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set Safety analysis set Safety analysis set Safety analysis set CTCAE Grade | Table 9.1 | Best Overall Response, Objective Response Rate, and Clinical Benefit Rate | Full analysis set |
| Adverse Events by System Organ Class and Preferred Term Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Safety analysis set Table 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set CTCAE Grade Safety analysis set CTCAE Grade Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set Safety analysis set | Table 9.2 | • | ECOG analysis set |
| Table 12 Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Safety analysis set Table 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set CTCAE Grade Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 10 | Adverse Events Overview | Safety analysis set |
| Table 13 Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set CTCAE Grade Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 11 | Adverse Events by System Organ Class and Preferred Term | Safety analysis set |
| Table 14 Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported Safety analysis set CTCAE Grade Table 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 12 | Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade | Safety analysis set |
| CTCAE Grade Fable 15.1 Adverse Events Leading to Carboplatin Discontinuation by Preferred Term Safety analysis set | Table 13 | Treatment-related Adverse Events by System Organ Class and Preferred Term | Safety analysis set |
| , , | Table 14 | · | Safety analysis set |
| Table 15.2Adverse Events Leading to Pemetrexed Discontinuation by Preferred TermSafety analysis set | Table 15.1 | Adverse Events Leading to Carboplatin Discontinuation by Preferred Term | Safety analysis set |
| | Table 15.2 | Adverse Events Leading to Pemetrexed Discontinuation by Preferred Term | Safety analysis set |

| Table 15.3 | Adverse Events Leading to OGX-427 Discontinuation by Preferred Term | Safety analysis set |
|---|---|---|
| Table 16.1 | Adverse Events Leading to Carboplatin Dose Reduction by Preferred Term | Safety analysis set |
| Table 16.2 | Adverse Events Leading to Pemetrexed Dose Reduction by Preferred Term | Safety analysis set |
| Table 16.3 | Adverse Events Leading to OGX-427 Dose Reduction by Preferred Term | Safety analysis set |
| Table 17 | Patient Deaths | All consented patients |
| Table 18.1 | Hematology CTCAE Grade Change from Baseline to Maximum on Treatment | Safety analysis set |
| Table 18.2 | Clinical chemistry CTCAE Grade Change from Baseline to Maximum on Treatment | Safety analysis set |
| Table 18.3 | Elevated AST, ALT, Total Bilirubin, and Alkaline Phosphate | Safety Analysis Set |
| Table 19 | Follow up Duration | Full analysis set |
| Table 20 | Serum Hsp27, Change from Baseline over Time | FAS with serum Hsp27 measurement |
| Figure 1.1 | Progression-free survival, Kaplan-Meier plot, Stratified by Arm | Full analysis Set |
| Figure 1.2 | Progression-free survival, Kaplan-Meier plot, Stratified by Arm and Baseline ECOG Performance | ECOG analysis Set |
| Figure 2.1 | Overall survival, Kaplan-Meier plot, Stratified by Arm | Full analysis Set |
| Figure 2.2 | Overall survival, Kaplan-Meier plot, Stratified by Arm and Baseline ECOG Performance | ECOG analysis Set |

Table 1 Patient Disposition All enrolleded patients

| | | Carboplatin<br>Pemetrexed | Carboplatin<br>Pemetrexed | |
|---|---|---|---|---|
| Disposition | Statistic | OGX-427 | Placebo | Total |
| Number of patients enrolled | n | | | xxx |
| Number of patients randomised | n | xx | XX | xxx |
| Number of patients un-treated | n | xx | xx | xxx |
| Number of patients treated | n | XX | XX | xxx |
| Number of patients with treatment discontinuation | n | xx | XX | xxx |
| Disease Progression | | XX | XX | XXX |
| RECIST | n | XX | XX | XXX |
| Clinical Progression | n | XX | XX | XXX |
| Adverse Event | n | XX | XX | XXX |
| Unable to complete at least 3 cycles of at least one chemotherapy agent | n | XX | XX | XXX |
| Patient requests to discontinue treatment | n | XX | XX | XXX |
| Patient requests to withdraw consent for the study | n | XX | XX | XXX |
| Non-compliance | n | XX | XX | XXX |
| Lost to follow-up | n | XX | XX | XXX |
| Death on study | n | XX | XX | XXX |
| Death due to disease progression | n | XX | XX | XXX |
| Death due to protocol therapy | n | XX | XX | xxx |
| Death due to AE<br>(Continued) | n | XX | XX | xxx |

Program Name: XXXX

## Table 1 Patient Disposition All consented patients

| isposition | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Death, cause unknown | n | XX | XX | XXX |
| Other | n | XX | XX | XXX |
| Other | n | XX | xx | XXX |

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

Table 2
Demographic Characteristics
Full analysis set

| Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| *************************************** | (/ | (/ | (=======) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX |
| Min | XX | XX | XX |
| Max | xx | xx | XX |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Mean | Pemetrexed OGX-427 Statistic (N=xx) n | Pemetrexed Pemetrexed Placebo Placebo |

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYYY)

Table 2
Demographic Characteristics
Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Demographic characteristic | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Asian | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <insert race=""></insert> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Ethnic group | | | | |
| Hispanic or Latino | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Non-hispanic or Latino | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| COG | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| obacco use | | | | |
| Smoker | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Non-Smoker | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x |

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYYY)

Table 3
Disease History
Full analysis set

| | 61 t t | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Patient characteristics | Statistic | (N=xx) | Pemetrexed | (N=xxx) |
| Histology | | | | |
| Adenocarcinoma | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Large Cell Carcinoma | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Stage at study entry | | | | |
| Stage IV at Initial Diagnosis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Recurrent Stage IV Disease | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| EGFR mutation status | | | | |
| Positive | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Negative | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ALK Translocation | | | | |
| Yes | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Fime from initial diagnosis to randomization (Months) [a] | | | | |
| N | n | XX | XX | XXX |
| Continued) | | | | |

<sup>[</sup>a] Month = (PHFPBDAT-PTRNDT+1)/30.4375.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Month = (PRGDAT-PTRNDT+1)/30.4375.

Table 3
Disease History
Full analysis set

| atient characteristics | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard deviation | SD | XX.XX | XX.XX | XX.XX |
| Median | Median | XX.X | XX.X | XX.X |
| Min | Min | XX.X | XX.X | XX.X |
| Max | Max | xx.x | XX.X | XX.X |
| | ation | | | |
| | ration<br>n | xx | xx | xxx |
| onths) [b] | | xx<br>xx.x | xx<br>xx.x | xxx<br>xx.x |
| | n | | | |
| N<br>Mean | n<br>Mean | XX.X | xx.x | xx.x |
| onths) [b] N Mean Standard deviation | n<br>Mean<br>SD | xx.x<br>xx.xx | xx.x<br>xx.xx | XX.X<br>XX.XX |

<sup>[</sup>a] Month = (PHFPBDAT-PTRNDT+1)/30.4375.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Month = (PRGDAT-PTRNDT+1)/30.4375.

Table 4
Prior Therapy
Full analysis set

| | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Prior systemic therapy | | | | |
| Missing | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Yes | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | n (%) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| Number of prior systemic regimens | | | | |
| 0 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 3 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Best overall response of prior systemic regimens [a] | | | | |
| Complete Response | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Partial Response | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Progressive Disease | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Stable Disease | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Not Evaluable | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Not Applicable | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Disease setting [a] | | | | |
| Neoadjuvant<br>(Continued) | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Patients with multiple categories or multiple times in a category will be tabulated one time in each category. Note: N/A = not applicable

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

Table 4 Prior Therapy Full analysis set

| | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Adjuvant | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| N/A | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Prior surgery | | | | |
| Missing | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Yes | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Prior radiotherapy | | | | |
| Missing | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Yes | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| No | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Patients with multiple categories or multiple times in a category will be tabulated one time in each category. Note: N/A = not applicable

Program Name: XXXX

Table 5.1

Laboratory Parameters at Baseline - Hematology

Full analysis set

| Hematology parameter | | | | | CTC | AE grade[a], | ૧ (%) | |
|---|---|---|---|---|---|---|---|---|
| | Arm | Treated,n | Randomized,n | G0 | G1 | G2 | G3 | G4 |
| Hemoglobin | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Placebo | xx | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Platelets | OGX-427 | xx | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Placebo | xx | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

[a] CTCAE = Common Terminology Criteria for Adverse Events (version 4.03).

Note: The number of randomized patients is the denominator for % calculation in each arm.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYYY)

Table 5.2

Laboratory Parameters at Baseline - Blood Chemistry

Full analysis set

| Blood chemistry parameter | | | | | CTC | CAE grade[a], | ૧ (%) | |
|---|---|---|---|---|---|---|---|---|
| | Arm | Treated,n | Randomized,n | G0 | G1 | G2 | G3 | G4 |
| Albumin | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Placebo | xx | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Glucose | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Placebo | XX | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<<pre><<parameter>>

[a] CTCAE = Common Terminology Criteria for Adverse Events (version 4.03).

Note: The number of randomized patients is the denominator for % calculation in each arm.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYYY)

 $\begin{tabular}{ll} Table 5.3 \\ Laboratory Parameters at Baseline - Liver Function Test \\ Full analysis set \end{tabular}$ 

| | | | | | CTC | AE grade[a], 1 | ૧ (%) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Liver function<br>parameter | Arm Treated, n Randomized, n | Treated,n Randomized,n | Arm Treated, n Randomized, n | rm Treated,n Randomized,n G0 G1 | Randomized,n | Randomized,n | G1 | G2 | G3 | G4 |
| SGPT/ALT | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| | Placebo | XX | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| SGOT/AST | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| | Placebo | XX | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| Alkaline Phosphatase | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| | Placebo | XX | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| Total bulirubin | OGX-427 | xx | xx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |
| | Placebo | XX | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | |

<sup>[</sup>a] CTCAE = Common Terminology Criteria for Adverse Events (version 4.03).

Note: The number of randomized patients is the denominator for % calculation in each arm.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYYY)

Table 6.1

Dose Exposure - Carboplatin

Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Parameter | Statistic | (N=XX) | (N=XX) | (N=xxx) |
| Total number of treatment cycles started | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 3 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 4 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Cumulative actual dose (AUC)[a] | | | | |
| n | n | X | X | X |
| Mean | Mean | xx.x | XX.X | XX.X |
| Standard Deviation | SD | XX.XX | XX.XX | xx.xx |
| Median | Median | XX.X | XX.X | XX.X |
| Minimum | Min | xx.x | XX.X | XX.X |
| Maximum | Max | xx.x | xx.x | XX.X |
| Duration (cycle)[b] | | | | |
| n | n | X | Х | x |
| Mean | Mean | XX.X | XX.X | XX.X |
| (Continued) | | | | |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by 6 multiplied by 100;

Table 6.1

Dose Exposure - Carboplatin

Full analysis set

| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total |
|---|---|---|---|---|
| Standard Deviation | SD | XX.XX | XX.XX | XX.XX |
| Median | Median | XX.X | XX.X | xx.x |
| Minimum | Min | XX.X | XX.X | XX.X |
| Maximum | Max | XX.X | xx.x | XX.X |
| Actual dose intensity (AUC/cycle)[c] | | | | |
| n | n | X | x | x |
| Mean | Mean | xx.x | XX.X | XX.X |
| Standard Deviation | SD | xx.xx | XX.XX | xx.xx |
| Median | Median | xx.x | XX.X | XX.X |
| Minimum | Min | xx.x | XX.X | XX.X |
| Maximum | Max | xx.x | xx.x | XX.X |
| Relative Dose Intensity (%)[d] | | | | |
| n | n | Х | X | X |
| Mean | Mean | xx.x | XX.X | XX.X |
| Standard Deviation | SD | XX.XX | XX.XX | XX.XX |
| Median | Median | XX.X | XX.X | xx.x |
| Minimum | Min | XX.X | XX.X | xx.x |
| (Continued) | | | | |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by 6 multiplied by 100;

SCRI Development Innovations

Protocol No.: LUN229

Page x of Y

### Table 6.1 Dose Exposure - Carboplatin Full analysis set

| | | Carboplatin<br>Pemetrexed | Carboplatin<br>Pemetrexed | |
|---|---|---|---|---|
| | | OGX-427 | Placebo | Total |
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Maximum | Max | xx.x | XX.X | XX.X |

[a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

- [c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.
- [d] Relative dose intensity is calculated as the actual dose intensity divided by 6 multiplied by 100;

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

Table 6.2

Dose Exposure - Pemetrexed

Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Total number of treatment phase cycles started | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 3 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 4 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total number of maintenance phase cycles started | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <insert number=""></insert> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Cumulative actual dose (mg/m2)[a] | | | | |
| n | n | X | X | x |
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard Deviation | SD | XX.XX | XX.XX | xx.xx |
| Median | Median | XX.X | XX.X | XX.X |
| Continued) | | | | |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by 500 multiplied by 100;

SCRI Development Innovations

Protocol No.: LUN229

Page x of Y

Table 6.2

Dose Exposure - Pemetrexed

Full analysis set

| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Minimum | Min | XX.X | XX.X | XX.X |
| Maximum | Max | xx.x | xx.x | XX.X |
| Duration (cycles)[b] | | | | |
| n | n | х | X | x |
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard Deviation | SD | xx.xx | XX.XX | xx.xx |
| Median | Median | XX.X | XX.X | XX.X |
| Minimum | Min | xx.x | XX.X | xx.x |
| Maximum | Max | xx.x | XX.X | XX.X |
| Actual dose intensity (mg/m2/cycle)[c] | | | | |
| n | n | X | x | X |
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard Deviation | SD | xx.xx | XX.XX | xx.xx |
| Median | Median | XX.X | XX.X | XX.X |
| Minimum | Min | XX.X | XX.X | XX.X |
| Maximum | Max | XX.X | XX.X | XX.X |

(Continued)

Program Name: XXXX

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by 500 multiplied by 100;

SCRI Development Innovations

Protocol No.: LUN229

Page x of Y

Table 6.2

Dose Exposure - Pemetrexed

Full analysis set

| Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| n | X | X | х |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min | XX.X | XX.X | xx.x |
| Max | XX.X | XX.X | XX.X |
| | n<br>Mean<br>SD<br>Median<br>Min | Pemetrexed | Pemetrexed Pemetrexed Placebo |

[a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

 ${\tt Datasets}\,({\tt date}): \ {\tt X\_XXX.XX}, \ {\tt X\_XXX.XXX} \ ({\tt DDMMMYYYYY})$ 

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/21.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by 500 multiplied by 100;

Table 6.3

Dose Exposure- OGX-427 or Placebo

Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Parameter | Statistic | (N=XX) | (N=xx) | (N=xxx) |
| Number of loading dose | | | | |
| 0 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 3 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Number of treatment phase cycles started | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 3 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 4 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Number of maintenance phase cycles started | | | | |
| 0 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 1 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 2 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <insert number=""></insert> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| (Continued) | | | | |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/7.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by the planned dose intensity multiplied by 100;

Table 6.3

Dose Exposure- OGX-427 or Placebo

Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Cumulative actual dose (mg)[a] | | | | |
| n | n | X | X | X |
| Mean | Mean | xx.x | XX.X | xx.x |
| Standard Deviation | SD | xx.xx | XX.XX | xx.xx |
| Median | Median | xx.x | XX.X | xx.x |
| Minimum | Min | xx.x | XX.X | xx.x |
| Maximum | Max | XX.X | XX.X | XX.X |
| Duration (weeks)[b] | | | | |
| n | n | x | X | x |
| Mean | Mean | xx.x | XX.X | xx.x |
| Standard Deviation | SD | xx.xx | XX.XX | xx.xx |
| Median | Median | xx.x | XX.X | xx.x |
| Minimum | Min | xx.x | xx.x | xx.x |
| Maximum | Max | XX.X | XX.X | XX.X |
| Actual dose intensity (mg/week)[c] | | | | |
| n | n | Х | Х | Х |
| (Continued) | | | | |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/7.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by the planned dose intensity multiplied by 100;

SCRI Development Innovations

Protocol No.: LUN229

Page x of Y

Table 6.3

Dose Exposure- OGX-427 or Placebo

Full analysis set

| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total (N=xxx) |
|---|---|---|---|---|
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard Deviation | SD | XX.XX | XX.XX | xx.xx |
| Median | Median | XX.X | XX.X | XX.X |
| Minimum | Min | XX.X | XX.X | xx.x |
| Maximum | Max | xx.x | xx.x | xx.x |
| Relative Dose Intensity (%)[d] | | | | |
| n | n | Х | X | x |
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard Deviation | SD | XX.XX | XX.XX | xx.xx |
| Median | Median | xx.x | XX.X | XX.X |
| Minimum | Min | XX.X | XX.X | XX.X |
| Maximum | Max | XX.X | XX.X | XX.X |

<sup>[</sup>a] Cumulative actual dose is the sum of the actual daily dose received from cycle 1 day 1 through treatment discontinue.

Program Name: XXXX

<sup>[</sup>b] Duration is calculated as the (last dose date - first dose date +1)/7.

<sup>[</sup>c] Actual dose intensity is calculated as the cumulative actual dose divided by the duration.

<sup>[</sup>d] Relative dose intensity is calculated as the actual dose intensity divided by the planned dose intensity multiplied by 100;

Table 6.4

Treatment Modifications - Carboplatin

Full analysis set

| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| | | , | , | , |
| Dose reduced | | | | |
| None | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 1 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 3 or more | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Infusion stopped/interrupted | | | | |
| None | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 1 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 2 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 3 or more | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Dose omitted/held | | | | |
| None | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 1 | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 2 | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Patients with 3 or more | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Discontinued | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Program Name: XXXX

Table 6.5
Treatment Modifications - Pemetrexed
Full analysis set

| Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| | , | , | , , |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | n(%) | Pemetrexed OGX-427 (N=xx) n(%) | Pemetrexed OGX-427 (N=xx) Pemetrexed Placebo (N=xx) n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) |

Program Name: XXXX
Table 6.6

Treatment Modifications - OGX-427 or Placebo
Full analysis set

| Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| n (웅) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | n(%) | Pemetrexed OGX-427 | Pemetrexed OGX-427 (N=xx) Pemetrexed Placebo (N=xx) n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) |

Program Name: XXXX

Table 7.1
Progression-free Survival
Full analysis set

| Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|------------------------------------------------|------------------|
| xx (xx.x) | xx(xx.x) |
| xx (xx.x) | xx (xx.x) |
| xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| xx) | |
| X | ) |

(Continued)

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

Note: Progression-free survival (PFS) is defined as the time from the date of radomization until the date of disease progression

(RECIST or clinical) or death due to any cause. Patients who have neither progression nor death will be censored.

Note: CI = Confidence Interval

Note: RECIST1.1

Program Name: XXXX

Datasets (date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

<sup>[</sup>b] The logrank test.

## Table 7.1 Progression-free Survival Full analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| p-values[b] | | | | |
| OGX-427 vs Placebo | p-value | x.xxxx | | |

[b] The logrank test.

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

Note: Progression-free survival (PFS) is defined as the time from the date of radomization until the date of disease progression

(RECIST or clinical) or death due to any cause. Patients who have neither progression nor death will be censored.

Note: CI = Confidence Interval

Note: RECIST1.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

| | | | <pre>Baseline ECOG Performance = 0</pre> | | Performance ≥ 1<br>xxx) |
|---|---|---|---|---|---|
| Parameter | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) |
| Number of patients progressed or died | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Number of patients censored | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Progression-free survival (PFS) [a], mont | hs | | | | |
| Median (95% CI) | Median (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 25th Percentile (95% CI) | 25th Percentile (95% C | I) xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 75th Percentile (95% CI) | 75th Percentile (95% C | I) xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| Event Rate [a], % | | | | | |
| 6 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 12 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |

(Continued)

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

Note: Progression-free survival (PFS) is defined as the time from the date of radomization until the date of disease progression (RECIST or clinical) or death due to any cause. Patients who have neither progression nor death will be censored.

Note: CI = Confidence Interval

Note: RECIST1.1

Program Name: XXXX

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

<sup>[</sup>b] The logrank test.

| | | <pre>Baseline ECOG Performance = 0</pre> | | <pre>Baseline ECOG Performance = 1</pre> | |
|---|---|---|---|---|---|
| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) |
| Hazard Ratio (two-sided 95% CI) | | , | | <u> </u> | |
| OGX-427 vs Placebo | x.xxx(x.xxx,x.xxx) | x.xxx(x.xxx,x.xxx) | | x.xxx(x.xxx,x.xxx) | |
| p-values[b] | | | | | |
| OGX-427 vs Placebo | p-value | x.xxxx | | x.xxxx | |

[b] The logrank test.

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

 ${\tt Note: Progression-free \ survival \ (PFS) \ is \ defined \ as \ the \ time \ from \ the \ date \ of \ radomization \ until \ the \ date \ of \ disease \ progression}$ 

(RECIST or clinical) or death due to any cause. Patients who have neither progression nor death will be censored.

Note: CI = Confidence Interval

Note: RECIST1.1

Program Name: XXXX

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

Table 8.1 Overall Survival Full analysis set

| | | Carboplatin | Carboplatin | |
|---|---|---|---|---|
| | | Pemetrexed | Pemetrexed | |
| | | OGX-427 | Placebo | Total |
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Number of patients died | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Number of patients censored | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Overall survival (OS) [a], months | | | | |
| Median (95% CI) | Median (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| 25th Percentile (95% CI) | 25th Percentile (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| 75th Percentile (95% CI) | 75th Percentile (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| Event Rate [a], % | | | | |
| 6 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| 12 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x |
| Hazard Ratio (two-sided 95% CI) | | | | |
| OGX-427 vs Placebo | x.xxx(x.xxx,x.xxx) | x.xxx(x.xxx,x.xxx) | | |
| n | | | | |

p-values[b]
(Continued)

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

Note: Overall survival (OS) is defined as the time from the date of randomization until the date of death due to any cause.

Note: CI = Confidence Interval

Program Name: XXXX

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

<sup>[</sup>b] The logrank test.

## Table 8.1 Overall Survival Full analysis set

| | | Carboplatin | Carboplatin | |
|--------------------|-----------|-------------|-------------|---------|
| | | Pemetrexed | Pemetrexed | |
| | | OGX-427 | Placebo | Total |
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| OGX-427 vs Placebo | p-value | x.xxxx | | |

\_\_\_\_\_\_

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: Overall survival (OS) is defined as the time from the date of randomization until the date of death due to any cause. Note: CI = Confidence Interval

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

<sup>[</sup>b] The logrank test.

| Parameter | | | Performance = 0<br>xxx) | <pre>Baseline ECOG Performance &gt;=</pre> | |
|---|---|---|---|---|---|
| | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) |
| Number of patients died | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Number of patients censored | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Overall survival (OS) [a], months | | | | | |
| Median (95% CI) | Median (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 25th Percentile (95% CI) | 25th Percentile (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 75th Percentile (95% CI) | 75th Percentile (95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| Event Rate [a], % | | | | | |
| 6 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| 12 months (95% CI) | Prob.(95% CI) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) | xx.x(xx.x, xx.x) |
| Hazard Ratio (one-sided 80% CI) | | | | | |
| OGX-427 vs Placebo (Continued) | x.xxx(x.xxx) | x.xxx(x.xxx) | | x.xxx(x.xxx) | |

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: Overall survival (OS) is defined as the time from the date of randomization until the date of death due to any cause.

Note: CI = Confidence Interval

Program Name: XXXX

 ${\tt Datasets}\,({\tt date}): \ {\tt X\_XXX.XX}, \ {\tt X\_XXX.XXX} \ ({\tt DDMMMYYYYY})$ 

<sup>[</sup>b] The logrank test.

Table 8.2
Overall Survival - Stratified by Baseline ECOG Performance
ECOG analysis set

| | | <pre>Baseline ECOG Performance = 0</pre> | | Baseline ECOG Performance $\geq$ 1 (N=xxx) | |
|---|---|---|---|---|---|
| Parameter | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) |
| Hazard Ratio (two-sided 95% CI)<br>OGX-427 vs Placebo | x.xxx(x.xxx,x.xxx) | x.xxx(x.xxx,x.xxx) | | x.xxx(x.xxx,x.xxx) | |
| p-values[b]<br>OGX-427 vs Placebo | p-value | x.xxx | | x.xxx | |

<sup>[</sup>a] Calculated using the Kaplan-Meier technique.

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: Overall survival (OS) is defined as the time from the date of randomization until the date of death due to any cause. Note: CI = Confidence Interval

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] The logrank test.

Table 9.1
Best Overall Response, Objective Response Rate, and Clinical Benefit Rate
Full analysis set

| Statistic n(%) n(%) | OGX-427<br>(N=xx)<br>xx(xx.x) | Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| n(%) | xx (xx.x) | , | (iv mm) |
| | | vv (vv v) | |
| n (%) | | AA (AA•A) | xx(xx.x) |
| ( 0 / | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| %, % | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| 용 (용,용) | | | xx.x(xx.x, xx.x) |
| p-value | | | X.XXXX |
| | n(%) n(%) n(%) n(%) n(%) n(%) %, % | n(%) xx(xx.x) n(%) xx(xx.x) n(%) xx(xx.x) n(%) xx(xx.x) n(%) xx(xx.x) xx(xx.x) xx(xx.x) xx(xx.x) xx(xx.x) xx(xx.x) xx(xx.x) | n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) n(%) xx(xx.x) xx(xx.x) %, % xx.x, xx.x xx.x, xx.x %(%,%) xx(xx.x) xx.x, xx.x |

(Continued)

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: CI = Confident Interval

- [a] Two sided exact 95% CI using the method of Clopper Pearson.
- [b] Fisher's exact test.

Program Name: XXXX

Table 9.1
Best Overall Response, Objective Response Rate, and Clinical Benefit Rate
Full analysis set

| | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Clinical benefit rate (CR+PR+SD≥months, CBR) | | , | , | |
| CBR | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 95% CI[a] | ે, ે | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Odds Ratio for CBR (two-sided 95% CI) | | | | |
| OGX-427 vs Placebo | 응 (응 <b>,</b> 응) | | | xx.x(xx.x, xx.x |
| p-value for CBR[b] | | | | |
| OGX-427 vs Placebo | p-value | | | x.xxxx |

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm.

Note: CI = Confident Interval

- [a] Two sided exact 95% CI using the method of Clopper Pearson.
- [b] Fisher's exact test.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

Table 9.2

Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG Performance

ECOG analysis set

| | Statistic | Baseline ECOG Po<br>(N=x: | | Baseline ECOG P<br>(N=x | |
|---|---|---|---|---|---|
| | | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) |
| Complete response (CR) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Partial response (PR) | n (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| Stable disease (SD months) | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Stable disease (SD<6 months) | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Progressive disease (PD) | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Clinical progression | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| RECIST progression | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Not evaluable (NE) | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Objective response rate (CR+PR, ORR) | | | | | |
| ORR | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 95% CI[a] | ુ, % | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Odds Ratio for ORR (two-sided 95% CI) | | | | | |
| OGX-427 vs Placebo<br>(Continued) | % (%, %) | xx.x(xx.x, xx.x) | | xx.x(xx.x, xx.x) | |

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: CI = Confident Interval

Program Name: XXXX

<sup>[</sup>a] Two sided exact 95% CI using the method of Clopper Pearson.

<sup>[</sup>b] Fisher's exact test.

Table 9.2

Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Stratified by Baseline ECOG Performance

ECOG analysis set

| | | Baseline ECOG Pe<br>(N=xx | | Baseline ECOG P (N=) | |
|---|---|---|---|---|---|
| | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) |
| p-value for ORR[b] | | | | | |
| OGX-427 vs Placebo | p-value | x.xxxx | | x.xxx | |
| Clinical benefit rate (CR+PR+SD months, | CBR) | | | | |
| CBR | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 95% CI[a] | %, % | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Odds Ratio for CBR (two-sided 95% CI) | | | | | |
| OGX-427 vs Placebo | 응 (응, 응) | xx.x(xx.x, xx.x) | | xx.x(xx.x, xx.x) | |
| p-value for CBR[b] | | | | | |
| OGX-427 vs Placebo | p-value | x.xxxx | | x.xxxx | |

Note: The denominator for the percentage calculation is the total number of patients who were assigned to the specific arm. Note: CI = Confident Interval

- [a] Two sided exact 95% CI using the method of Clopper Pearson.
- [b] Fisher's exact test.

Program Name: XXXX

 ${\tt Datasets (date): X\_XXX.XX, X\_XXX.XXX \ (DDMMMYYYYY)}$ 

Table 10
Adverse Events Overview
Safety analysis set

| | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with at least one: | | | | |
| Adverse event | | | | |
| Grade 1 / Mild | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 2 / Moderate | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 3 / Severe | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 4 / Life Threatening | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 5 / Fatal | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Treatment-related adverse event | | | | |
| Grade 1 / Mild | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 2 / Moderate | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 3 / Severe | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 4 / Life Threatening | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Grade 5 / Fatal | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Serious adverse event | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Treatment-related serious adverse event | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Serious adverse event leading to death<br>Continued) | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Patients with multiple events in the same category are counted only once in that category.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03).

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

Table 10
Adverse Events Overview
Safety analysis set

| | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| | Statistic | (N=xx) | | |
| reatment-related serious adverse event leading to death | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| dverse events leading to treatment discontinued | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| dverse events leading to treatment stopped/interrupted | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| dverse events leading to treatment omitted/held | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| dverse events leading to treatment reduced | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

[a] Patients with multiple events in the same category are counted only once in that category.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03).

Program Name: XXXX

Table 11

Adverse Events by System Organ Class and Preferred Term

Safety analysis set

| edDRA system organ class | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|
| Preferred term | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| atients with any AE [a] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| nfections and infestations | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ervous system disorders | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Headache | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Dizziness | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| insert System organ class> | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

[a] Number (%) of patients with AEs, sorted on international order for system organ class and alphabetical order for preferred term Note: A patient can have one or more preferred terms reported under a given system organ class.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Table 12

Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade

Safety analysis set

| MedDRA system organ class | Maximum | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|---|
| Preferred term | CTCAE grade | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| Patients with any AE [a] | Total | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 4 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 5 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Infections and infestations | Total | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n (웅) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 4 | n (웅) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 5 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Respiratory tract infection NOS | Total | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Continued) | | | | | |

<sup>[</sup>a] Each patient has only been represented with the maximum reported CTCAE grade for each system organ class / preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03)

Program Name: XXXX

Number (%) of patients with AEs, sorted by international SOC order and alphabetical PT and then maximum grade.

 ${\tt Table~12}$  Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade Safety analysis set

| MedDRA system organ class Preferred term | Maximum<br>CTCAE grade | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|
| | 4 | n (%) | x (xx.x) | x (xx.x) | x (xx.x) |
| | 5 | n (%) | x(xx.x) | x(xx.x) | x(xx.x) |

<insert Preferred term>

[a] Each patient has only been represented with the maximum reported CTCAE grade for each system organ class / preferred term.

Number (%) of patients with AEs, sorted by international SOC order and alphabetical PT and then maximum grade.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03)

Program Name: XXXX

Table 13

Treatment-related Adverse Events by System Organ Class and Preferred Term Safety analysis set

| MedDRA system organ class<br>Preferred term | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| | | (2) 2222/ | (=: ====, | (2: 22222) |
| Patients with any treatment-related AE [a] | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Infections and infestations | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ervous system disorders | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Headache | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Dizziness | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Kinsert System organ class> | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

<sup>[</sup>a] Number (%) of patients with AEs, sorted on international order for system organ class and alphabetical order for preferred term Note: A patient can have one or more preferred terms reported under a given system organ class.

Table 14

Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade

Safety analysis set

| | | | Carboplatin<br>Pemetrexed | Carboplatin<br>Pemetrexed | |
|---|---|---|---|---|---|
| MedDRA system organ class Preferred term | Maximum | Statistic | OGX-427<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xxx) |
| Fieleffed term | CTCAE grade | Statistic | (N-XX) | (N-XX) | (IV-XXX) |
| Patients with any treatment-related AE [a] | Total | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 4 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 5 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Infections and infestations | Total | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 4 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 5 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Respiratory tract infection NOS | Total | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | 1 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 2 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 3 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Continued) | | | | | |

<sup>[</sup>a] Each patient has only been represented with the maximum reported CTCAE grade for each system organ class / preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03)

Program Name: XXXX

Number (%) of patients with AEs, sorted by international SOC order and alphabetical PT and then maximum grade.

Table 14

Treatment-related Adverse Events by System Organ Class, Preferred Term and Maximum Reported CTCAE Grade

Safety analysis set

| MedDRA system organ class | Maximum . | | Carboplatin<br>Pemetrexed<br>OGX-427 | Carboplatin<br>Pemetrexed<br>Placebo | Total |
|---|---|---|---|---|---|
| Preferred term | CTCAE grade | Statistic | (N=xx) | (N=xx) | (N=xxx) |
| | 4 | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| | 5 | n (%) | x(xx.x) | x(xx.x) | x(xx.x) |

<insert Preferred term>

[a] Each patient has only been represented with the maximum reported CTCAE grade for each system organ class / preferred term.

Number (%) of patients with AEs, sorted by international SOC order and alphabetical PT and then maximum grade.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Note: CTCAE = Common Terminology Criteria for Adverse Events (version 4.03)

Program Name: XXXX

Table 15.1

Adverse Events Leading to Carboplatin Discontinuation by Preferred Term

Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to Carboplatin dose discontinuation [a] [b] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Number (%) of patients with an AE leading to discontinuation of Carboplatin, sorted by alphabetically for preferred term.

Patients with multiple AEs leading to discontinuation are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Action taken, Carboplatin discontinued.

Table 15.2

Adverse Events Leading to Pemetrexed Discontinuation by Preferred Term

Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to Pemetrexed dose discontinuation [a] [b] | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Number (%) of patients with an AE leading to discontinuation of Pemetrexed, sorted by alphabetically for preferred term. Patients with multiple AEs leading to discontinuation are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Action taken, Pemetrexed discontinued.

Table 15.3

Adverse Events Leading to OGX-427 Discontinuation by Preferred Term

Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to OGX-427 dose discontinuation [a] [b] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Number (%) of patients with an AE leading to discontinuation of OGX-427, sorted by alphabetically for preferred term.

Patients with multiple AEs leading to discontinuation are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Action taken, OGX-427 discontinued.

Table 16.1

Adverse Events Leading to Carboplatin Dose Reduction by Preferred Term

Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to Carboplatin dose reduction [a] [b] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

 $<sup>\</sup>hbox{[a] Number (\$) of patients with an AE leading to reduction of Carboplatin, sorted by alphabetically for preferred term.}\\$ 

Patients with multiple AEs leading to reduction are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Action taken, Carboplatin reduced.

 ${\bf Table~16.2}$  Adverse Events Leading to Pemetrexed Dose Reduction by Preferred Term Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to Pemetrexed dose reduction [a] [b] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Number (%) of patients with an AE leading to reduction of Pemetrexed, sorted by alphabetically for preferred term.

Patients with multiple AEs leading to reduction are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYYY)

<sup>[</sup>b] Action taken, Pemetrexed reduced.

Table 16.3

Adverse Events Leading to OGX-427 Dose Reduction by Preferred Term

Safety analysis set

| MedDRA Preferred term | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Patients with any AE leading to OGX-427 dose reduction [a] [b] | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Respiratory tract infection NOS | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pharyngitis | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Influenza | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <pre><insert preferred="" term=""></insert></pre> | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

<sup>[</sup>a] Number (%) of patients with an AE leading to reduction of OGX-427, sorted by alphabetically for preferred term.

Patients with multiple AEs leading to reduction are counted once for each preferred term.

Note: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of study treatment.

Note: MedDRA version 17.1

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>b] Action taken, OGX-427 reduced.

Table 17
Patient Deaths
All enrolled patients

| Category | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Total number of alive | n (%) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| Total number of deaths | n (%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Death due to disease progression | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Death due to protocol therapy | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Death due to AE | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Death, cause unknown | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Other | n(%) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Note: Rows are mutually exclusive, patients are only reported in one category.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYYY)

 ${\small \textbf{Table 18.1}}$  Hematology CTCAE Grade Change from Baseline to Maximum on Treatment Safety analysis set

| | | | | Maximum overall CTCAE grade during treatment (%)[c] | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Hematology<br>Variable | Arm | | Patients at baseline[b] n(%) | Grade 0<br>n(%) | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total<br>n(%) |
| Hemoglobin | OGX-427 (N=xx) | 0 | x (x.x) | x(x.x) | x (x.x) | x(x.x) | x (x.x) | x(x.x) | xx(x.x) |
| | 0011 127 (11 1111) | 1 | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 2 | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 3 | x (x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 4 | x(x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x(x.x) | xx (x.x) |
| | | Total evaluable | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) |
| | Placebo (N=xx) | 0 | x(x.x) | x(x.x) | x (x.x) | x (x.x) | x(x.x) | x (x.x) | xx(x.x) |
| | | 1 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 2 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 3 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 4 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | Total evaluable | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) |

<<Variable >>

Note: CTCAE Common Terminology Criteria for Adverse Events version 4.03.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

<sup>[</sup>a] Baseline is defined as the last result obtained prior to the start of study treatment

<sup>[</sup>b] Patients with a baseline value and at least one on-treatment value. Percentages have been calculated using the number of patients with a baseline value and a post baseline value.

<sup>[</sup>c] Derived from laboratory assessments between the start of treatment and 30 days following the date of last dose of study medication and is the maximum CTCAE grade.

Table 18.2
Clinical chemistry CTCAE Grade Change from Baseline to Maximum on Treatment
Safety analysis set

| | | | | Maximum overall CTCAE grade during treatment (%)[c] | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Hematology<br>Variable | Arm | Baseline CTCAE<br>grade[a] | Patients at baseline[b] n(%) | Grade 0<br>n(%) | Grade 1 | Grade 2<br>n(%) | Grade 3 n(%) | Grade 4 | Total<br>n(%) |
| Albumin | OGX-427 (N=xx) | 0 | x (x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x(x.x) | xx (x.x) |
| | (4. 1111, | 1 | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 2 | x (x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 3 | x (x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | xx (x.x) |
| | | 4 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | Total evaluable | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) |
| | Placebo (N=xx) | 0 | x (x.x) | x(x.x) | x (x.x) | x (x.x) | x (x.x) | x(x.x) | xx (x.x) |
| | | 1 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 2 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 3 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | 4 | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | x(x.x) | xx(x.x) |
| | | Total evaluable | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) | xx(x.x) |

<<Variable >>

Note: CTCAE Common Terminology Criteria for Adverse Events version 4.03.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

<sup>[</sup>a] Baseline is defined as the last result obtained prior to the start of study treatment

<sup>[</sup>b] Patients with a baseline value and at least one on-treatment value. Percentages have been calculated using the number of patients with a baseline value and a post baseline value.

<sup>[</sup>c] Derived from laboratory assessments between the start of treatment and 30 days following the date of last dose of study medication and is the maximum CTCAE grade.

Table 18.3
Elevated AST, ALT, Total Bilirubin, and Alkaline Phosphate
Safety analysis eet

| Parameter Abnormality | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| AST | | | | |
| N N | n(%) | x(xx.x) | x (xx.x) | x (xx.x) |
| 3x - <5x ULN | n(%) | x (xx.x) | x (xx.x) | x (xx.x) |
| 5x - <10x ULN | n(%) | x (xx.x) | x (xx.x) | x (xx.x) |
| 10x - <20x ULN | n(%) | x (xx.x) | x (xx.x) | x (xx.x) |
| >=20x ULN | n (%) | x (xx.x) | x (xx.x) | x (xx.x) |
| ALT | | | | |
| N | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 3x - <5x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 5x - <10x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 10x - <20x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| >=20x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| AST or ALT | | | | |
| N | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 3x - <5x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 5x - <10x ULN | n (%) | x(xx.x) | x(xx.x) | x(xx.x) |
| 10x - <20x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| >=20x ULN<br>Continued) | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |

Note: ULN = upper limit of normal; AST = Aspartate transaminase; ALT = Alanine transaminase; Tbili = Total Bilirubin.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

Table 18.3
Elevated AST, ALT, Total Bilirubin, and Alkaline Phosphate
Safety analysis eet

| Parameter Abnormality | Statistic | Carboplatin Pemetrexed OGX-427 (N=xx) | Carboplatin Pemetrexed Placebo (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| ratameter Aphormaticy | Statistic | (N-XX) | (IV-XX) | (IV-XXX) |
| Total Bilirubin | | | | |
| N | n (%) | x(xx.x) | x(xx.x) | x(xx.x) |
| >2x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| Alkaline Phosphatase | | | | |
| N | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| >1.5x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| (AST or ALT) and Total Bilirubin | | | | |
| N | n(%) | x (xx.x) | x(xx.x) | x(xx.x) |
| (AST or ALT $>3x$ ULN ) and $2x$ ULN $>$ Tbili $>$ 1.5x ULN | n(%) | x(xx.x) | x(xx.x) | x(xx.x) |
| (AST or ALT $>3x$ ULN ) and Tbili $>= 2x$ ULN | n (%) | x(xx.x) | x(xx.x) | x(xx.x) |

Note: ULN = upper limit of normal; AST = Aspartate transaminase; ALT = Alanine transaminase; Tbili = Total Bilirubin.

Program Name: XXXX

Table 19 Follow up Duration Full analysis set

| | Statistic | Carboplatin<br>Pemetrexed<br>OGX-427<br>(N=xx) | Carboplatin<br>Pemetrexed<br>Placebo<br>(N=xx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| ollow up duration (months) | | | | |
| n | n | xx | XX | XX |
| Mean | Mean | XX.X | XX.X | XX.X |
| Standard deviation | SD | xx.xx | XX.XX | XX.XX |
| Median | Median | xx | XX | XX |
| Min | Min | xx | XX | XX |
| Max | Max | xx | XX | XX |

Program Name: XXXX

Table 20 Serum Hsp27, Change from Baseline over Time FAS with serum Hsp27 measurement

| | | | Observed Results | | | | % Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Protocol Timepoint | N | Mean | SD | Min | Median | Max | N | Mean | SD | Min | Median | Max |
| OGX427 (N=xx) | Pre-treatment | XX | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | | | | | | |
| | Pre-loading dose | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX | | | | | | |
| | Cycle 1 day 1 | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX | XX | XX.XX | XX.XXX | xx.xx | XX.XX | XX.XX |
| | Cycle n day 1 | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX | XX | XX.XX | XX.XXX | xx.xx | XX.XX | XX.XX |
| | End of Treatment | XX | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx | XX | XX.XX | xx.xxx | xx.xx | XX.XX | XX.XX |
| Placebo (N=xx) | Pre-treatment | XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | | | | | | |
| | Pre-loading dose | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX | | | | | | |
| | Cycle 1 day 1 | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX |
| | Cycle n day 1 | XX | xx.xx | XX.XXX | XX.XX | XX.XX | XX.XX | XX | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XX |
| | End of Treatment | XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX | xx.xx | xx.xxx | XX.XX | XX.XX | XX.XX |

Note: Baseline is defined as the last value observed before the administration of study treatment.

Note: % Change from baseline = 100\* (related protocol timepoint value - baseline value)/(baseline value).

Program Name: XXXX

 ${\tt Datasets (date): X\_XXX.XX, X\_XXX.XXX \ (DDMMMYYYYY)}$ 

Figure 1.1 Progression-free survival, Kaplan-Meier plot, Stratified by Arm Full analysis Set



Note: + indicates a censored observation.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

 $Figure \ 1.2 \\ Progression-free \ survival, \ Kaplan-Meier plot, \ Stratified \ by \ Arm \ and \ Baseline \ ECOG \ Performance \\ ECOG \ analysis \ Set$ 



Note: + indicates a censored observation.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)

Figure 2.1

Overall survival, Kaplan-Meier plot, Stratified by Arm

Full analysis Set



Note: + indicates a censored observation.

Program Name: XXXX

Datasets(date): X\_XXX.XX, X\_XXX.XXX (DDMMMYYYY)

Figure 2.2

Overall survival, Kaplan-Meier plot, Stratified by Arm and Baseline ECOG Performance ECOG analysis Set



Note: + indicates a censored observation.

Program Name: XXXX

Datasets(date): X XXX.XX, X XXX.XXX (DDMMMYYYY)